CLINICAL TRIAL: NCT03858335
Title: Therapeutic Effects of Constraint-Induced Movement Therapy on Young Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Yi Kwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-06-100-008
Record Dates: First submitted 2019-02-25; First posted 2019-02-28 (Actual); Results first posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Cerebral Palsy Spastic Hemiplegic
Keywords: constraint-induced movement therapy; hemiplegia; hand function; gross motor
MeSH Terms: conditions — Hemiplegia | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Constraint-induced movement therapy (Experimental): Children in constraint-induced movement therapy (CIMT) group will wear forearm splint on the unaffected arm 24 hours for 3 weeks, and receive 15 mCIMT sessions(30-hour dosage)
  Interventions: Other: Constraint-induced movement therapy
- Control (No Intervention): Children in control group will receive only traditional rehab therapies without wearing splint

INTERVENTIONS:
Other: Constraint-induced movement therapy — The constraint-induced movement therapy (CIMT) program requires children to wear forearm splint on the unaffected arm 24 hours for 3 weeks. The program consists of 5 sessions per week for 3 weeks.
  Arms: Constraint-induced movement therapy

SUMMARY:
This study evaluates the therapeutic effects of constraint-induced movement therapy on infants and children with hemiplegic cerebral palsy. Half of the participants will receive CIMT (constraint-induced movement therapy) and others will not.

DETAILED DESCRIPTION:
This study evaluates the therapeutic effects of constraint-induced movement therapy on infants and children with hemiplegic cerebral palsy. Half of the participants will receive CIMT (constraint-induced movement therapy) and others will not.

Participants will be randomly assigned to either CIMT group or control group. Children of the CIMT group will wear forearm splint 24 hours for 3 weeks to inhibit use of the unaffected arm.

ELIGIBILITY:
Inclusion Criteria:

* spastic hemiplegic cerebral palsy patients
* 7~36 months old

Exclusion Criteria:

* cognitive impairment severe enough to make participation impossible
* uncontrolled epilepsy
* visual or hearing impairment
* musculoskeletal disorders

Ages: 7 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2019-09-28 (Actual); Study Completion 2019-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Yi Kwon, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Constraint-induced Movement Therapy | Control
Started | 16 | 16
Completed | 12 | 12
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Constraint-induced Movement Therapy | Control | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 15.9 (8.4) | 17.3 (6.2) | 16.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 12 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Pediatric Motor Activity Log (PMAL) Score at Post Test
Description: The PMAL was derived from the Motor Activity Log, which is used as an assessment tool in adults who participated CIMT, to measure changes in upper extremity use in real life. This parental assessment tool rates the use of the children's affected upper extremities in daily activities. Twenty-two arm-hand functional tasks that are typical for children aged 7 months to 8 years (e.g., taking off socks or shoes, holding a cup) were assessed and collected as a systemic data. The test has two components: (1) how often (PMAL HO) and (2) how well (PMAL HW). Parents rate PMAL HO on a 6-point scale from 0 (not at all) to 5 (all the time) and PMAL HW from 0 (does not use) to 5 (same as the unaffected arm). This tool has a high test-retest reliability (r=0.94; P<0.01) and a high internal consistency (Cronbach's α=0.88 to 0.95).
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Constraint-induced Movement Therapy | Control
Number analyzed (Participants) | 12 | 12
score on a scale
  how well | 0.83 (0.58) | 0.00 (0.57)
  how often | 0.50 (0.35) | -0.05 (0.56)

2. Primary Outcome: Change From Baseline Accelerometers_Vector Magnitude Average Counts(VMA) at Post Test
Description: To evaluate the upper limb use in the real-world, participants wore two accelerometers (one on each wrist). Three variables were measured using accelerometers: vector magnitude average counts (VMA), percent of time in moderate to vigorous physical activity (% MVPA), and use ratio (UR). VMA refers to the magnitude of the resulting vector that forms when combining the sampled acceleration from all three axes.
Time Frame: baseline and 4 weeks
Population: Only children who agreed to participate in the accelerometer study(n=8) wore accelerometers.
Measure: Mean (Standard Deviation); unit: counts per minute
Arm/Group | Constraint-induced Movement Therapy | Control
Number analyzed (Participants) | 4 | 4
counts per minute | 44.73 (12.8) | 8.78 (14.94)

3. Secondary Outcome: Change From Baseline Pediatric Evaluation of Disability Inventory (PEDI) at Post Test
Description: The Pediatric Evaluation of Disability Inventory (PEDI) is a reliable and valid parent-report assessment that evaluates the performance, changes, and capabilities of functional activities in children with disabilities aged between 6 months and 7.5 years. Within the three domains of (1) self-care, (2) mobility, and (3) social function, it measures three scales: (1) functional skills; (2) caregiver assistance; and (3) modifications. In this study, only the functional skills scale was used because it directly evaluates the current capabilities of selected tasks. Therefore, the PEDI scores in this study reflect the functional skill of the children on a scale between 0 and 100: 0 indicates no ability, and 100 indicates full capability to perform the selected items.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Constraint-induced Movement Therapy | Control
Number analyzed (Participants) | 12 | 12
score on a scale
  self-care | 2.25 (2.30) | 1.25 (1.48)
  mobility | 2.83 (1.64) | 2.83 (4.67)
  social function | 2.83 (3.27) | 0.75 (0.75)

4. Secondary Outcome: Change From Baseline Peabody Developmental Motor Scales-2 (PDMS-2) at Post Test
Description: The PDMS-2 is a standardized, norm-referenced test, which includes gross motor and fine motor domains. All items of the PDMS-2 are scored on a 3-point scale (0 to 2): 0 is assigned when the child cannot perform the item or when the attempts do not meet the criteria of the item; 1 is assigned when the attempts do not meet for successful performance, but the behavior is emerging; and 2 indicates that the behavior is emerging, and the criterion for successful performance is fully met. The standard score and developmental age equivalent are obtained by converting the raw score of each subtest according to the criteria of the PDMS-2 manual; the standard score was used for this study. The interrater reliability and internal consistency of the fine motor domain were reported as 0.98 and 0.96, respectively. The predictive validity was reported as 0.91.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Constraint-induced Movement Therapy | Control
Number analyzed (Participants) | 12 | 12
score on a scale
  grasping | 0.83 (1.80) | -0.83 (2.89)
  visual motor integration | 0.92 (1.24) | -0.67 (1.61)

5. Secondary Outcome: Change From Baseline Gross Motor Function Measure (GMFM) at Post Test
Description: GMFM-88 is a measure developed to evaluate the gross motor function changes in CP children. It has five components: lying and rolling, sitting, kneeling and crawling, standing, and walking. The score of each dimension is expressed as a percentage of the maximum score. The GMFM-66, which includes 66 items of the original 88 items. Item scoring is the same for the GMFM-88 and the GMFM-66. There is a scoring system with each item scored as 0, 1, 2, 3, or "not tested". A scoring key of 0 - does not initiate, 1 - initiates, 2 - partially completes, and 3 - completed, is used. Scoring the GMFM-66 requires the use of a computer program called the Gross Motor Ability Estimator (GMAE). Individual item scores are entered and a mathematical algorithm calculates an interval level total score. The total score is an estimate of the child's gross motor function. The range of total score is from 0 to 100. The higher values represent a better outcome.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Constraint-induced Movement Therapy | Control
Number analyzed (Participants) | 12 | 12
score on a scale | 3.33 (2.55) | 4.37 (2.37)

6. Secondary Outcome: Change From Baseline Accelerometers_% Moderate to Vigorous Physical Activity(MVPA) at Post Test
Description: MVPA is a category of activity intensity, which is measured with metabolic equivalents (METs). Moderate-intensity physical activity is defined as 3-6 METs, and vigorous-intensity physical activity is defined as any activity above 6 METs. This means that MVPA is any activity over 3 METs.
Time Frame: baseline and 4 weeks
Population: Only children who agreed to participate in the accelerometer study(n=8) wore accelerometers.
Measure: Mean (Standard Deviation); unit: percentage of moderate to vigorous PA
Arm/Group | Constraint-induced Movement Therapy | Control
Number analyzed (Participants) | 4 | 4
percentage of moderate to vigorous PA | -2.67 (0.91) | 0.51 (1.31)

7. Secondary Outcome: Change From Baseline Accelerometers_Use Ratio at Post Test
Description: Use Ratio was calculated by dividing the hours of use of the affected limb by the hours of use of the non-affected limb (affected use/unaffected use).
Time Frame: baseline and 4 weeks
Population: Only children who agreed to participate in the accelerometer study(n=8) wore accelerometers.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Constraint-induced Movement Therapy | Control
Number analyzed (Participants) | 4 | 4
Ratio | 0.01 (0.01) | -0.02 (0.07)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Continuous restraint could be harsh on infants and toddlers because they are too young. Therefore, this study used detachable splints, not casts, in children in the CIMT group to allow them to detach it during washes and before sleeping. In addition, considering that adverse events such as increase in stress/crying, sleep disorders, or skin rashes could occur, we asked their parents to detach the splints and report if any of those problems had occurred.
Arm/Group | Constraint-induced Movement Therapy | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT03858335/Prot_SAP_000.pdf